CLINICAL TRIAL: NCT05836480
Title: Immediate Suboptimal Result of Mitral Valve Repair: Late Implications in a Matched Cohort Study
Status: Completed | Type: Observational
Sponsor: Michele De Bonis (Other)
Responsible Party: Sponsor-Investigator, Michele De Bonis, Chief of Cardiac Surgery of Advance and Research Therapies, Ospedale San Raffaele
Organization: Ospedale San Raffaele (Other)
Other Study IDs: SUB-MVR
Record Dates: First submitted 2023-01-27; First posted 2023-05-01 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Mitral Regurgitation
MeSH Terms: conditions — Mitral Valve Insufficiency | interventions — Mitral Valve Annuloplasty

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Suboptimal repair: Patients discharged with a residual mitral regurgitation of at least moderate (2+)degree
  Interventions: Procedure: mitral valve repair
- Optimal repair: Patients discharged with a residual mitral regurgitation of mild (1+) or less degree (trace or 0)
  Interventions: Procedure: mitral valve repair

INTERVENTIONS:
Procedure: mitral valve repair — conservative surgery to treat mitral regurgitation. A mitral valve plasty is performed according to the most appropriate technique

SUMMARY:
Mitral valve regurgitation is a pathology affecting the left atrioventricular valve, conditioning the loss of the normal unidirectionality of the atrioventricular flow and therefore volumetric and pressure overload of the left heart chambers. In industrialized countries, the most common etiology of mitral regurgitation is degenerative mitral disease.

Mitral valve repair surgery represents the gold standard for the treatment of severe degenerative mitral regurgitation. The expected optimal result would be the absence of residual post-procedural mitral regurgitation, even if it is not uncommon to obtain a valve with residual regurgitation of a mild degree. In some cases, for various reasons (technical difficulties, long aortic clamping time, advanced age, high pre-operative surgical risk), a suboptimal result is accepted, i.e. a post-procedural residual mitral regurgitation of even a moderate degree ( 0, 1+, or 2+/4+).

The aim of the present study is to evaluate the late clinical and echocardiographic implications of suboptimal mitral valve repair with a paired-data cohort study

ELIGIBILITY:
Inclusion Criteria:

* Study group:
* presence of severe degenerative mitral regurgitation treated by mitral valve repair between 2006 and 2013;
* presence of moderate residual mitral regurgitation at discharge.
* Control group:
* presence of severe degenerative mitral regurgitation treated by mitral valve repair between 2006 and 2013;
* presence of residual mitral regurgitation of at least mild grade at discharge.

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent surgical mitral valve repair. Patients of study (Suboptimal) group were discharged with a 2+ or more residual mitral regurgitation, patients in control group (Optimal) were discharged with a 1+ or less residual mitral regurgitation
Sampling Method: Non-Probability Sample
Enrollment: 141 (Actual)
Dates: Start 2019-10-05 (Actual); Primary Completion 2019-10-15 (Actual); Study Completion 2019-10-15 (Actual)

PRIMARY OUTCOMES:
Mortality | through study completion, a minimum of 6 years

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Ospedale San Raffaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: No